CLINICAL TRIAL: NCT06030427
Title: A Virtual Mindfulness and Weight Management Program for Those With Cancer Histories to Mitigate Risk of Relapse and Improve Wellbeing: A Feasibility Study
Brief Title: Virtual Mindfulness and Weight Management to Mitigate Risk of Relapse and Improve Wellbeing in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-004890; NCI-2023-06407 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-004890 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2024-11

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods; Health Promotion; Interviews as Topic; Mindfulness; Mindfulness-Based Stress Reduction; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (virtual mindfulness and weight management) (Experimental): Patients participate in a virtual behavioral weight management program with an integrated mindfulness component consisting of 12, 75-minute virtual group sessions over 12 weeks to help improve mood, coping strategies, stress management, and weight loss. Patents also receive patient education handouts, view behavioral educational PowerPoint presentations over 30 minutes, and wear a Fitbit on study.
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Educational Intervention; Other: Health Promotion and Education; Other: Internet-Based Intervention; Other: Interview; Other: Medical Device Usage and Evaluation; Behavioral: Mindfulness Relaxation; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Participate in weight management program
Other: Educational Intervention — Receive patient education handouts
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Health Promotion and Education — View behavioral educational PowerPoint presentation
Other: Internet-Based Intervention — Complete virtual behavioral weight management with an integrated mindfulness component program
Other: Interview — Ancillary studies
Other: Medical Device Usage and Evaluation — Wear Fitbit
Behavioral: Mindfulness Relaxation — Complete mindfulness components
  Other Names: MBSR; Mindful Meditation; Mindfulness Meditation; Mindfulness-Based Stress Reduction
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well a virtual mindfulness and weight management program to mitigate risk of relapse and improve well being for obese cancer survivors in community practice and rural areas. Obesity has been linked to increased risk for certain kinds of cancer and is the second highest modifiable risk factor for cancer. It is also well documented that having a cancer diagnosis and treatment is a stressful experience. It is hoped that an addition of a 10-minute mindfulness-based stress reduction exercise to the virtual positive health habits group focused on weight management can improve wellbeing and distress. Virtual care options continue to extend the reach of medical providers to cancer survivors, particularly those in the rural setting. A virtual behavioral weight management program with an integrated mindfulness component may improve mood, coping strategies, stress management, and weight loss among community practice and rural obese cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess if a 12-week virtual weight management program with a mindfulness component will improve well-being of obese cancer patients with a specific focus on self-reported measures of depression and anxiety.

II. To assess if a mindfulness component added to the virtual behavioral weight management will promote weight loss, improve mood, and increase physical activity.

OUTLINE:

Patients participate in a virtual behavioral weight management program with an integrated mindfulness component consisting of 12, 75-minute virtual group sessions over 12 weeks to help improve mood, coping strategies, stress management, and weight loss. Patents also receive patient education handouts, view behavioral educational PowerPoint presentations over 30 minutes, and wear a Fitbit on study.

ELIGIBILITY:
Inclusion Criteria:

* 18 or over
* Identified stage I, II, or III cancer in remission
* Body mass index (BMI) of 30 or greater
* English as a primary language
* Has access to a device with a camera (computer, tablet, or video capable phone) that has wifi and reliable internet access

Exclusion Criteria:

* Unable to provide consent
* Eastern Cooperative Oncology Group (ECOG) performance status scale score of 3 or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
General anxiety disorder-7 (GAD-7) | Baseline; 12 weeks
  Assessed by change in GAD-7 scores from a total score for seven items ranges from 0 to 21: 0-4 (minimal anxiety); 5-9 (mild anxiety); 10-14 (moderate anxiety); 15-21 (severe anxiety).
Patient Health Questionnaire (PHQ)-8 | Baseline; 12 weeks
  Assessed by change in PHQ-8 scores, as measured by a total score of 4 items from 0-12: 0-2 (normal); 3-5 (mild depression); 6-8 (moderate depression); 9-12 (severe depression).
Feasibility of virtual mindfulness and weight management program | 12 weeks
  Assessed by the extent to which participants adhere to the intervention. Will be quantified based on number of sessions attended out of a possible 12.

SECONDARY OUTCOMES:
Body weight | Baseline; 12 weeks
  Assessed by change in body weight
Body composition parameter | Baseline; 12 weeks
  Will be assessed in a fasted state or 3 hour post meal by subjects standing on a scale without socks or shoes.
Daily activity levels - heart rate | Baseline; 12 weeks
  Will be assessed by heart rate monitoring as recorded by a wrist-worn accelerometer (Fitbit Inspire)
Daily activity levels - activity | Baseline; 12 weeks
  Will be assessed from data recorded by a wrist-worn accelerometer monitoring fitness activity.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Howell, Ph.D., Principal Investigator — Mayo Clinic Health System-Franciscan Healthcare
Locations (1):
- Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials